CLINICAL TRIAL: NCT06383312
Title: Investigation of the Effectiveness of Reflexologic Magnetic Insoles on Dysmenorrhea Symptoms in Primary Dysmenorrhea
Brief Title: Magnetic Reflexologic Insoles for Primary Dysmenorrhea
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, gizem boztas, Assistant Professor, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-772.02-4248
Record Dates: First submitted 2024-04-06; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Primary Dysmenorrhea
Keywords: Dysmenorrhea; Reflexology; Pain; Foot Orthoses
MeSH Terms: conditions — Dysmenorrhea; Pain

STUDY DESIGN:
Intervention Model Description: two groups; treatment group and sham group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reflexologic Magnetic Insoles Group (Active Comparator): Participants will place the insoles inside their shoes and use them for at least 7 hours a day, every day, for 12 weeks.
  Interventions: Device: Reflexologic Magnetic Insole Group
- Orthopedic Insoles Group (Sham Comparator): Participants will place the insoles inside their shoes and use them for at least 7 hours a day, every day, for 12 weeks.
  Interventions: Device: Orthopedic Insole Group

INTERVENTIONS:
Device: Reflexologic Magnetic Insole Group — Reflexologic magnetic insole will be used for at least 7 hours a day, every day, for 12 weeks in participants diagnosed with primary dysmenorrhea. Then the effectiveness of the insoles will be compared.
  Arms: Reflexologic Magnetic Insoles Group
Device: Orthopedic Insole Group — Orthopedic insole (sham) will be used for at least 7 hours a day, every day, for 12 weeks in participants diagnosed with primary dysmenorrhea. Then the effectiveness of the insoles will be compared.
  Arms: Orthopedic Insoles Group

SUMMARY:
In the study, easy-to-access and easy-to-use reflexologic magnetic insoles were used in women with primary dysmenorrhea who did not want to receive medical treatment; In addition to reducing symptoms such as pain, nausea, dizziness, fainting, vomiting, weakness, constipation/acute gastroenteritis, it is aimed to increase individuals' participation in daily life activities and increase their quality of life by increasing their emotional state.

DETAILED DESCRIPTION:
60 women diagnosed with primary dysmenorrhea through examination by a gynecologist will be included in the study. 60 women will be randomly divided into 2 groups. These groups; Reflexologic Magnetic Insoles Sham Group: They will use orthopedic insoles.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with primary dysmenorrhea
* Visual Analogue Scale (VAS) value is 3 and above
* The patient has cooperation
* Having regular menstruation

Exclusion Criteria:

* Getting pregnant during treatment
* Using analgesic medication
* Visual Analogue Scale (VAS) value should be between 0-3
* Having pain in another part of the body

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Since dysmenorrhea is a problem seen in the menstrual cycle in women, female participants will be included in the study.
Enrollment: 60 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
McGill Pain Questionnaire-Short Form: | 12 weeks
  It evaluates the sensory dimension of pain and the affective dimension of pain. Affective and sensory dimension scores of pain are measured with a Likert-type scale (0-No pain, 3-Severe Pain). The total pain dimension subparametric is the sum of the sensory dimension and the affective dimension of the pain. Total pain intensity is measured with a 6-point Likert-type scale (0-No pain, 5-Unbearable Pain). A high score indicates a high level of pain.
Menstruation Attitude Questionnaire | 12 weeks
  Valuated subdimensions include menstruation as a deliberating event, menstruating as a bothersome event, menstruation as a natural event, anticipation and prediction of the onset of menstruation, and denial of any effects of menstruation. The scale is evaluated with a 5-point Likert-type." A high mean score indicates a "positive" attitude toward menstruation.
Menstruation Symptom Questionnaire | 12 weeks
  It contains 24 items. It is a 5-point Likert type scale. Participants are asked to evaluate the symptoms that occur during menstruation as a-never (1), b-rarely (2), c-sometimes (3), d-often (4) and e-always (5). The overall score of the scale is calculated by taking the average of the total score obtained from the scale items. A higher score indicates that the symptoms are experienced more clearly.
Visual Analogue Scale (VAS) | 12 weeks
  The Visual Analogue Scale (VAS) is used to convert non-numerical values to digital. The value 0 means I have no pain, 10 means I have unbearable pain. The person marks his pain on this ruler. It measures the intensity of the pain.

CONTACTS AND LOCATIONS:
Overall Officials: Gizem BOZTAŞ ELVERİŞLİ, Ph.D, Study Director — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No